CLINICAL TRIAL: NCT02478905
Title: TransFLUas: Transmission of Influenza Virus From Asymptomatic Healthcare Workers and Inpatients in the Acute Care Hospital Setting: A Prospective Study Over Two Consecutive Influenza Seasons
Brief Title: Transmission of Influenza Virus From Asymptomatic Healthcare Workers and Inpatients in the Acute Care Hospital Setting
Acronym: TransFLUas
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Schweizerischer Nationalfonds (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2015-0228
Record Dates: First submitted 2015-06-05; First posted 2015-06-23 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Human Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Virological analyses
  * Influenza A and B PCR from nasal swabs
  * Whole genome sequencing of positive swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- surveillance cohort: Flocked mid-turbinate nasal swabs for influenza PCR will be collected from study participants daily
  Interventions: Other: Influenza

INTERVENTIONS:
Other: Influenza

SUMMARY:
The epidemiology and transmission dynamics of influenza in hospitals are only poorly understood, particularly with respect to subjects without symptoms of influenza infection (e.g. without fever, cough, sore throat, nasal congestion, weakness, headache, loss of appetite, or myalgia). Knowledge about whether asymptomatic subjects are able to transmit influenza is of major importance. If they do transmit influenza, vaccination of patients and healthcare workers (HCW) before start of the influenza season, the permanent use of masks by HCW during influenza season, and quarantine for previously exposed inpatients may be the only available measures to reduce the number of influenza transmission events from asymptomatic subjects in acute care hospitals. Closure of this knowledge gap would be of major benefit to infection prevention and control recommendations, and may in turn reduce morbidity and mortality associated with influenza in hospitals through improved patient management.

DETAILED DESCRIPTION:
The epidemiology and transmission dynamics of influenza in hospitals are only poorly understood, particularly with respect to subjects without symptoms of influenza infection (e.g. without fever, cough, sore throat, nasal congestion, weakness, headache, loss of appetite, or myalgia). Knowledge about whether asymptomatic subjects are able to transmit influenza is of major importance. If they do transmit influenza, vaccination of patients and healthcare workers (HCW) before start of the influenza season, the permanent use of masks by HCW during influenza season, and quarantine for previously exposed inpatients may be the only available measures to reduce the number of influenza transmission events from asymptomatic subjects in acute care hospitals.

The investigators' key aim is therefore to define whether exposure to asymptomatic subjects with influenza infection constitutes a risk for influenza transmission in an acute care hospital setting through active, prospective surveillance.

The investigators' secondary aims are to describe the prevalence of community-acquired symptomatic and asymptomatic influenza upon hospital admission and the incidence of asymptomatic and symptomatic nosocomial influenza among inpatients; to assess transmission dynamics of symptomatic influenza infection in acute care; and to study the incidence of asymptomatic and symptomatic influenza, absenteeism (i.e. being absent from work due to influenza), presenteeism (i.e. being present at work despite influenza infection) associated with influenza, and compliance with infection control recommendations to prevent spread of influenza in acute care HCW.

The investigators plan to enroll 1,260 inpatients and 180 HCW from medical wards at the University Hospital Zurich in a prospective study over two consecutive influenza seasons in order to detect at least one transmission event from an asymptomatic individual shedding influenza virus. Flocked mid-turbinate nasal swabs will be collected daily from consenting inpatients starting from day of admission until two days after discharge and from HCW over the influenza (winter) season and analyzed for influenza A and B using polymerase chain reaction. Simultaneously, signs and symptoms of influenza infection (including cough, sore throat, fever >37.8°C, nasal congestion, weakness, headache, loss of appetite or myalgia) as well as contact patterns between inpatients and HCW will be recorded. Reconstruction of influenza transmission chains will be based on phylogenetic analyses derived from next-generation sequence data and epidemiological contact tracing.

ELIGIBILITY:
Inclusion Criteria:

* 18 or more years of age;
* Available for follow-up during the study period;
* If a HCW: employed full- or part-time (≥50% full-time equivalent);
* Understand the study, agree to its provisions, and give written informed consent (as documented by signature).

Exclusion Criteria:

* If a HCW: planning to spend more than two consecutive weeks outside of Switzerland during the winter study period (November 1st to April 31st);
* If a HCW: planning to take leave from work for more than two consecutive weeks during the winter study period (e.g. maternity or medical leave);
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders or dementia of the subject;
* Known or suspected non-compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This project is a prospective study following patients in medical wards and acute care HCW (including nursing staff (nurses and assistant nurses), physiotherapists, house staff with direct patient contact and medical doctors (clinical fellows) working on the same wards at the University Hospital Zurich. Inpatients and HCW will be recruited from general medical and infectious diseases wards, pulmonology wards, hematology wards and from the stem cell transplant unit. All HCW and inpatients on the ward under surveillance are eligible for the study
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2016-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Secondary attack rate of asymptomatic or presymptomatic influenza among inpatients, among acute care workers and between inpatients and acute care HCW in an acute care hospital setting | up to 6 months
  diagnosed by positive influenza PCR from flocked mid-turbinate nasal swab collected in symptomatic or asymptomatic individuals following face-to-face contact with an individual with symptomatic influenza infection on the day of contact.

SECONDARY OUTCOMES:
Secondary attack rate of symptomatic influenza among inpatients, among acute care workers and between inpatients and acute care HCW in an acute care hospital setting | up to 6 months
  Secondary attack rate of symptomatic influenza among inpatients, among acute care workers and between inpatients and acute care HCW in an acute care hospital setting: as diagnosed by positive influenza PCR from flocked mid-turbinate nasal swab collected in symptomatic or asymptomatic individuals following face-to-face contact with an individual with symptomatic influenza infection on the day of contact. Transmissions will be considered 'proven' if confirmed by phylogenetic analyses. Specifically, we expect that whole-genome sequence analysis will demonstrate identical or almost identical influenza strains within transmission chains.
  Transmissions will be considered 'probable' if there is epidemiological evidence of face-to-face contact and identical strains have been identified in PCR but whole-genome sequencing was technically unsuccessful;
Proportion of asymptomatic and symptomatic inpatients with influenza infection upon hospital admission: as diagnosed by influenza polymerase chain reaction (PCR) from flocked mid-turbinate nasal swabs collected upon hospital admission | up to 6 months
  diagnosed by influenza PCR from flocked mid-turbinate nasal swabs collected upon hospital admission
Incidence of asymptomatic (A5) and symptomatic (A6) nosocomial influenza in hospital inpatients, defined as the number of emerging influenza infections >72 hours after hospital admissions per 100 patient-days | up to 6 months
  diagnosed by PCR from flocked mid-turbinate nasal swabs collected three times per week over the influenza season
Incidence of asymptomatic (A7) and symptomatic (A8) influenza in acute care hospital workers defined as the number of influenza infections per 100 HCW per influenza season | up to 6 months
  diagnosed by influenza PCR from flocked mid-turbinate nasal swabs collected three times per week over the influenza season collected three times per week over the influenza season
Association of individual influenza symptoms with influenza transmission from subjects with symptomatic influenza infection | up to 6 months
  Association of individual influenza symptoms with influenza transmission from subjects with symptomatic influenza infection
Influenza-attributable mortality in inpatients, expressed as infection-fatality rate, i.e. number of deaths among those infected | up to 6 months
  number of deaths among those infected
Absenteeism: as defined by total number of days absent from work due to PCR-proven influenza divided by total number of days due to work in HCW | up to 6 months
  Absenteeism: as defined by total number of days absent from work due to PCR-proven influenza divided by total number of days due to work in HCW;
Presenteeism: as defined by total number of days with symptoms of influenza present at work divided by total number of days due to work in HCW with PCR-proven influenza infection | up to 6 months
  Presenteeism: as defined by total number of days with symptoms of influenza present at work divided by total number of days due to work in HCW with PCR-proven influenza infection;
Compliance with hand hygiene recommendations and cough etiquette (including barrier precautions) in HCW according to repeated observations | up to 6 months
  Compliance with hand hygiene recommendations and cough etiquette (including barrier precautions) in HCW according to repeated observations;
Association of patient and HCW characteristics, including receipt of influenza vaccine, with asymptomatic viral shedding, as compared to symptomatic shedding | up to 6 months
  Association of patient and HCW characteristics, including receipt of influenza vaccine, with asymptomatic viral shedding, as compared to symptomatic shedding;
Association between viral load and asymptomatic or symptomatic transmission based on quantification of viral shedding according to cycle threshold (Ct) values from PCR | up to 6 months
  defined as the number of cycles required for the fluorescent signal to cross the threshold (i.e. exceeds background level).

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kuster, MD, Principal Investigator — Division of Infectious Diseases and Hospital Epidemiology
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Kuster SP, Boni J, Kouyos RD, Huber M, Schmutz S, Shah C, Bischoff-Ferrari HA, Distler O, Battegay E, Giovanoli P, Guckenberger M, Kohler M, Muller R, Petry H, Ruschitzka F, McGeer A, Coleman BL, Sax H, Weber R, Trkola A. Absenteeism and presenteeism in healthcare workers due to respiratory illness. Infect Control Hosp Epidemiol. 2021 Mar;42(3):268-273. doi: 10.1017/ice.2020.444. Epub 2020 Nov 26. PMID 33239124
- [Derived] Schwarz H, Boni J, Kouyos RD, Turk T, Battegay E, Kohler M, Muller R, Petry H, Sax H, Weber R, McGeer A, Trkola A, Kuster SP. The TransFLUas influenza transmission study in acute healthcare - recruitment rates and protocol adherence in healthcare workers and inpatients. BMC Infect Dis. 2019 May 21;19(1):446. doi: 10.1186/s12879-019-4057-5. PMID 31113375